CLINICAL TRIAL: NCT02268929
Title: Integrated Personalized Diabetes Management (Integrated PDM):Prospective, Randomized, Controlled Intervention Study for the Evaluation of the Effectiveness and the Benefit of Integrated PDM in the Care of People With Type 2 Diabetes in General Medical Practices in Germany (GP).
Brief Title: A German Study Evaluating the Efficacy and the Benefit of Integrated Personalized Diabetes Management (PDM) for Type 2 Diabetes Patients.
Acronym: PDM-ProValueGP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RD001231
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2017-11-24 (Actual); Status verified 2017-11

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): Patients treated by usual customary medical practice (Usual Care)
  Interventions: Device: Accu-Chek Smart Pix readout Device
- Intervention Group (Other): Patients treated with "Integrated Personalized Diabetes Management"
  Interventions: Device: Accu-Chek Smart Pix Software

INTERVENTIONS:
Device: Accu-Chek Smart Pix Software — Software with adherence evaluation software used according to Integrated Personalized Diabetes Management (PDM)
  Arms: Intervention Group
Device: Accu-Chek Smart Pix readout Device — Smartpix device for data upload out from blood glucose meter devices
  Arms: Control Group

SUMMARY:
This study is a German, prospective, multicenter, controlled, cluster-randomized, interventional comparative study evaluating the efficacy and benefits of integrated PDM care by measuring HbA1c levels in patients with Type 2 Diabetes. Patients will be randomized into two groups to use Accu-Chek Smartpix software and Accu-Chek Smartpix device.

DETAILED DESCRIPTION:
Outcome of both studies (RD001732 and RD001231) will be integrated and additionally reported as PDM-ProValue study program (Integrated Personalized Diabetes Management) due to the high similarity in study characteristics, design and study results.

ELIGIBILITY:
Inclusion Criteria:

* Existence of a signed Informed Consent form (before any study procedure)
* Diagnosed Type 2 diabetes mellitus
* Age =18 years
* Insulin therapy for =6 months: BOT, SIT, CT or ICT
* HbA1c =7.5% within the last 6 weeks before study visit 1 (patient's inclusion)
* Longer-term diabetes care by the trial site (at least for the duration of the 12-month study participation)
* General practitioner is the primary practitioner in the diabetes care of the patient
* Insured by the statutory health insurance (GKV) as a statutory or voluntarily insured member or as a family co-insured member
* Willing and able to participate in the study and to follow the study procedures, among other things sufficient command of the German language, spoken and written

Exclusion Criteria:

* Diabetes treatment by insulin pump therapy (CSII)
* Experience with the use of special software for systematic processing of SMBG data, e.g. the Accu-Chek® Smart Pix System/Software, the Accu-Chek® 360° Software and/or the Diabetes Software DIABASS
* Presence of terminal renal failure / dialysis and/or a loss of sight or a tumor illness
* Chronic use of steroids in adrenal suppressant doses, of other immuno-modulatory drugs or chemotherapy
* Known alcohol, drug and medication abuse
* Known metabolic disorders and/or disorders or therapies that could lead to or have led to wrong measured results (e.g. with the blood glucose measurement)
* Existing pregnancy, breast-feeding or plan to become pregnant during study participation
* Physical illness and/or psychological disorder with the result that the patient cannot implement the medical treatment recommendations independently
* Dependency relationship to the sponsor or to the investigator, e.g. as a professional colleague or family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2014-10-14 (Actual); Primary Completion 2017-01-11 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
The mean HbA1c change by Generalized Estimating Equations (GEE) methods | from Baseline to 12 months

SECONDARY OUTCOMES:
Effects of integrated Personalized Diabetes Management (PDM) by means of Generalized Estimating Equations [GEE] methods | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Iris Vesper, Study Director — Roche Diabetes Care
Locations (46):
- Germany (46):
  - Albstadt
  - Auerbach/Vogtland
  - Bad Kreuznach
  - Beucha
  - Beutel/Templin
  - Blankenhain
  - Bochum
  - Bockenem
  - Borna
  - Bremerhaven
  - Cloppenburg
  - Dransfeld
  - Dresden
  - Düren
  - Elsterwerda
  - Essen
  - Föhren
  - Geringswalde
  - Giessen
  - Hanover
  - Hemsbach
  - Herborn
  - Kerpen
  - Köthen
  - Krefeld
  - Kreuzau
  - Leipzig
  - Löhne
  - Lübeck
  - Mainz
  - Meissen
  - Meudt
  - Papenburg
  - Reinfeld
  - Riesa
  - Rochlitz
  - Rodgau
  - Schleiden
  - Schwedt
  - Schweich
  - Siegen
  - Sigmaringen
  - Staufenberg
  - Trier
  - Weida
  - Wetzlar